CLINICAL TRIAL: NCT07307196
Title: THE EFFECT OF A MİNDFULNESS-BASED STRESS REDUCTİON PROGRAM ON PREGNANCY ADAPTATİON, STRESS, AND FETAL ANXİETY LEVELS İN WOMEN WHO CONCEİVED AFTER INFERTİLİTY TREATMENT: A RANDOMİZED CONTROLLED TRİAL
Brief Title: The Effect of a Mindfulness-Based Stress Reduction Program on Pregnancy Adaptation, Stress, and Fetal Anxiety Levels in Women Who Conceived After Infertility Treatment
Acronym: MBSR-PAFS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kahramanmaras Sutcu Imam University (Other)
Responsible Party: Principal Investigator, Hatice Gul OZTAS, DR., Kahramanmaras Sutcu Imam University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: KahramanmaraşSIUI9
Record Dates: First submitted 2025-12-13; First posted 2025-12-29 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Infertile Females or Females With Ovarian Insufficiency; Pre - Delivery Pregnant Women
Keywords: infertility; pregnancy; stress; midwifery
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): MBSRParticipants allocated to the experimental arm will receive a structured Mindfulness-Based Stress Reduction (MBSR) program in addition to routine prenatal care. The MBSR intervention is delivered in a group format by a trained researcher and is adapted for pregnant women who conceived following infertility treatment. The program is conducted over 4 weeks, with two sessions per week.
  Each session includes guided mindfulness practices such as breathing-focused meditation, body scan exercises, gentle pregnancy-safe yoga movements, emotional awareness practices, and self-compassion exercises. The intervention also includes mindfulness practices aimed at strengthening maternal-fetal bonding, such as loving-kindness meditation directed toward the fetus and mindful awareness of bodily sensations related to pregnancy. Participants are encouraged to engage in daily home practice using provided audio-guided materials.
  The primary purpose of this arm is to reduce pregnancy-related stress a
  Interventions: Behavioral: MBSR
- control group (No Intervention): Participants allocated to the control arm will receive routine prenatal care only and will not participate in any structured mindfulness or psychological intervention during the study period. After completion of post-intervention assessments, participants in the control arm will be offered the MBSR program upon request.

INTERVENTIONS:
Behavioral: MBSR — Participants allocated to the experimental arm will receive a structured Mindfulness-Based Stress Reduction (MBSR) program in addition to routine prenatal care. The MBSR intervention is delivered in a group format by a trained researcher and is adapted for pregnant women who conceived following infertility treatment. The program is conducted over 4 weeks, with two sessions per week.
  Each session includes guided mindfulness practices such as breathing-focused meditation, body scan exercises, gentle pregnancy-safe yoga movements, emotional awareness practices, and self-compassion exercises. The intervention also includes mindfulness practices aimed at strengthening maternal-fetal bonding, such as loving-kindness meditation directed toward the fetus and mindful awareness of bodily sensations related to pregnancy. Participants are encouraged to engage in daily home practice using provided audio-guided materials.
  The primary purpose of this arm is to reduce pregnancy-related stress and fe
  Arms: Experimental

SUMMARY:
Infertility treatment is a long and challenging process. Women who become pregnant after this process may experience stress, anxiety and intense concerns about the baby's health alongside their happiness. These feelings can negatively affect the mother's adjustment to pregnancy and her psychological well-being.

This study was designed to examine the effects of the Mindfulness-Based Stress Reduction (MBSR) programme, administered to women who became pregnant after infertility treatment, on:

stress levels during pregnancy,

adaptation to pregnancy,

and foetal (baby's health-related) anxiety.

Pregnant women participating in the study will be divided into two groups: an experimental group and a control group. Women in the experimental group will receive mindfulness-based stress reduction training lasting approximately 4 weeks. This programme includes breathing exercises, meditation, body awareness, self-compassion exercises, and practices aimed at strengthening the mother-baby bond. The control group will not receive any training during this period.

Translated with DeepL.com (free version)

DETAILED DESCRIPTION:
Infertility treatment is a physically and emotionally demanding process. Although achieving pregnancy after infertility treatment is often perceived as a positive outcome, many women continue to experience significant psychological challenges during pregnancy, including heightened stress, difficulty adapting to pregnancy, and persistent anxiety regarding fetal health. These emotional responses may negatively affect maternal well-being, pregnancy adaptation, and pregnancy outcomes. Despite the growing body of evidence supporting mindfulness-based interventions during pregnancy, there is limited research focusing specifically on women who conceive following infertility treatment.

Mindfulness-Based Stress Reduction (MBSR) is a structured, evidence-based program that aims to enhance awareness of present-moment experiences through mindfulness practices such as meditation, breathing exercises, body awareness, gentle yoga, and self-compassion practices. Previous studies have demonstrated that MBSR can effectively reduce stress and anxiety and improve psychological well-being in various populations, including pregnant women and women undergoing infertility treatment. However, the effects of MBSR on pregnancy adaptation and fetal health anxiety among women who become pregnant after infertility treatment have not been adequately investigated.

This randomized controlled study is designed to evaluate the effectiveness of an MBSR program on pregnancy adaptation, perceived stress, and fetal health anxiety in women who conceived following infertility treatment. Eligible participants will be randomly assigned to either an intervention group or a control group. The intervention group will receive an MBSR program delivered over four weeks, consisting of structured sessions that include mindfulness meditation, breathing-focused practices, body scan exercises, gentle yoga, emotional awareness, self-compassion training, and practices aimed at strengthening maternal-fetal bonding. Participants will also be encouraged to engage in daily mindfulness practices at home.

The control group will receive routine prenatal care and will not participate in any structured psychological or mindfulness-based intervention during the study period. After completion of post-intervention assessments, participants in the control group who wish to receive the MBSR training will be offered the program.

Data will be collected at baseline (pre-test) and after completion of the intervention (post-test) using validated instruments to assess pregnancy-related distress, pregnancy adaptation, and fetal health anxiety. The primary outcomes of the study are changes in perceived stress levels, pregnancy adaptation, and fetal health anxiety scores between the intervention and control groups.

The findings of this study are expected to provide evidence on the potential benefits of MBSR as a supportive, non-pharmacological intervention for improving psychological well-being and pregnancy adaptation in women who conceive following infertility treatment. The results may contribute to the development of holistic, evidence-based prenatal care approaches and inform healthcare professionals about effective strategies to support this vulnerable population.

ELIGIBILITY:
Inclusion Criteria:

* As a result of infertility treatment,
* Pregnancy week 10-28. Pregnant women in their 10th to 28th week of pregnancy
* with no foetal abnormalities,
* without any psychiatric diagnosis,
* able to communicate and willing to participate in the study

Exclusion Criteria:

* Pregnant women who participated in mind-body practices or any prenatal class/programme during the study period.
* Those with communication difficulties

Min Age: 18 Months | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2026-01-10 (Estimated); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Tilburg Distress in Pregnancy Scale | 1 month
  Description: It was developed by Pop et al. in the Netherlands in 2011 for the diagnosis of distress in pregnancy. It was translated into Turkish by Çapık in 2013 after a Turkish validity and reliability study. The scale consists of a total of 16 items. It is 4-point Likert type. The lowest score that can be obtained from the total scale is 0 and the highest score is 48. The scale has two sub-dimensions as 'Negative affect' and 'Partner involvement'. The scale can be applied to pregnant women aged 12 weeks and above. Cronbach's alpha coefficient of the original scale was 0.78. The Cronbach's alpha coefficient of the Turkish form of the scale is 0.80 (Çapık et al. 2015).
Prenatal Self-Assessment Scale (PSAS) | 1 month
  Developed by Lederman in 1979 to assess adaptation to motherhood (Lederman 1979), the validity and reliability of this scale in Turkish were established in 2006 by Beydağ and Mete in 21 health centres in the province of Denizli. This four-point Likert-type scale consists of 79 items. The scale has seven subscales: thoughts about one's own and the baby's health, acceptance of pregnancy, acceptance of the maternal role, readiness for childbirth, fear of childbirth, relationship with one's own mother, and relationship with one's spouse. Each subscale contains between 10 and 15 items (Beydağ and Mete 2008). Forty-seven of the items in this scale are reverse-scored (1, 2, 3, 4, 6, 7, 8, 10, 11, 12, 14, 15, 18, 19, 20, 21, 22, 23, 24, 25, 26, 28, 31, 32, 33, 35, 37, 38, 40, 47, 48, 49, 50, 53, 55, 56, 59, 60, 61, 70, 71, 72, 73, 74, 75, 78, 79) (Beydağ and Mete 2008). Each item on the scale
  Translated with DeepL.com (free version)
Fetal Anxiety Scale (FAS) | 1 month
  The scale, developed by Reiser and Wright (2019), measures pregnant women's anxiety about the health of their foetus. The FAS has no subscales and consists of 14 items. Each item consists of 4 statements that best reflect the experiences of pregnant women in the past weeks. Items on the scale are scored from 0 (no symptoms) to 3 (severe symptoms), and the sum of the items yields the total foetal health anxiety score (0-42), with higher scores indicating increased levels of foetal health anxiety. The scale's Cronbach's alpha value is 0.85 (Gökbulut et al., 2024).

CONTACTS AND LOCATIONS:
Locations (1):
- Kahramanmaraş Sütçü İmama Universty, Kahramanmaraş, K.maraş, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No